CLINICAL TRIAL: NCT06776588
Title: Study on the Diagnosis of Ground-glass Lung Cancer by Microwave Ablation Combined With Puncture Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beidahuang Industry Group General Hospital (Other)
Responsible Party: Principal Investigator, LiuMingyang, Director, Beidahuang Industry Group General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Golden staff
Record Dates: First submitted 2024-11-18; First posted 2025-01-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation combined with biopsy (Experimental): Microwave ablation combined with biopsy
  Interventions: Procedure: Microwave ablation combined with biopsy

INTERVENTIONS:
Procedure: Microwave ablation combined with biopsy — CT thin-layer scanning 3D reconstruction is used, and AI and fragment omics technology are used to evaluate the risk of malignant transformation of pulmonary nodules. Microwave ablation of pulmonary nodules is combined with intraoperative rapid pathology technology to determine the nature of punctured tissue and the degree of ablation, and to explore the optimal ablation time and ablation power.

SUMMARY:
This study is a multicenter study. It plans to screen 200 patients with pulmonary nodule lesions with ground glass as the main body, take CT thin-layer scanning 3D reconstruction, apply AI and fragment omics technology to evaluate the risk of malignant transformation of pulmonary nodules, and use microwave ablation to treat pulmonary nodules and combine intraoperative rapid pathology technology to determine the nature of puncture tissue and the degree of ablation, and then explore the optimal ablation time and ablation power.

DETAILED DESCRIPTION:
Combining AI and fragmentomics technology, this study enrolled 200 patients with ground-glass lung cancer for comprehensive evaluation. By collecting detailed characteristic data of ground-glass lung cancer, including nodule diameter, average CT value, solid component ratio (CTR), nodule morphology and other related signs, CT imaging and AI technology, and fragmentomics technology were used for comprehensive analysis to form a set of joint strategies to efficiently screen and diagnose patients with early lung cancer.

Microwave ablation is used to treat lung nodules, and intraoperative rapid pathology technology is used to determine the nature of the punctured tissue and the degree of ablation (observing pathological changes in the lesion area, including cancer cell death and fibrosis of the lesion tissue), determine whether the lesion has been completely ablated, or whether there are residual active cancer cells, and then explore the optimal ablation time and ablation power.

Finally, long-term follow-up of patients after microwave ablation, including collection of intraoperative/postoperative complication data, regular CT review, evaluation of treatment effect, monitoring for recurrence, and improving individualized treatment plans for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 75 years;
2. GGN patients with the maximum axial diameter of the lesion in the lung window ≤ 3 cm;
3. Refusing radical surgery or being unable to tolerate surgical treatment;
4. Normal coagulation function, platelet count ≥ 60 × 109 /L;
5. ECOG score ≤ 2 points;

Exclusion Criteria:

1. Patients with the maximum axial diameter of the lesion in the lung window greater than 3 cm
2. Platelets <50×109 /L
3. Patients with severe bleeding tendency and coagulation dysfunction that cannot be corrected in the short term
4. Severe chronic obstructive pulmonary disease, emphysema, pulmonary fibrosis and pulmonary hypertension
5. Patients whose anticoagulant therapy or antiplatelet drugs have been discontinued for less than 5 days before ablation
6. Patients with severe heart, liver, kidney and brain dysfunction
7. Patients with severe anemia, dehydration and cachexia that cannot be corrected or improved in the short term
8. Patients with an estimated survival period of less than 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Local contral rate | up to 36 months
  LCR is the rate of CR, PR plus SD
Recurrence-free survival | up to 36 months
  It estimates the recurrence-free rate of patients who have already survived, with no history of metastasis, a certain period of time.
Overall Survival | up to 36 months
  Defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Detection rate | up to 36 months
  The detection rate of early lung cancer was calculated

OTHER OUTCOMES:
To explore the optimal ablation time | up to 36 months
  To explore the optimal ablation time
To explore the optimal power selection | up to 36 months
  To explore the optimal power selection

CONTACTS AND LOCATIONS:
Locations (1):
- Beidahuang Industry Group General Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No